CLINICAL TRIAL: NCT07143448
Title: Phase Ib, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study Assessing the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of HS235 Added to Background Treatment in Adults With PAH
Brief Title: A Study of HS235 for Treatment of Pulmonary Arterial Hypertension (PAH) in Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 35Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS235-002
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HS235 (Experimental): HS235 Subcutaneous Injection
  Interventions: Biological: HS235
- Placebo (Placebo Comparator): Subcutaneous Injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HS235 — Subcutaneous Injection
  Arms: HS235
Other: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
Phase 1b Study of HS235 Assessing the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of the Activin Signaling Inhibitor HS235 Added to Background Treatment in Adults with Pulmonary Arterial Hypertension (PAH)

DETAILED DESCRIPTION:
A Phase Ib, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study Assessing the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of the Activin Signaling Inhibitor HS235 Added to Background Treatment in Adults with Pulmonary Arterial Hypertension (PAH)

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if they meet all of the following criteria:

1. Male and female patients, 18 years of age and older.
2. Body Mass Index (BMI) 18.5 and 40 kg/m2 and body weight at or below 120 kg.
3. Baseline Right Heart Catheterization (RHC) performed during the Screening Period documenting minimum pulmonary vascular resistance (PVR) of ≥ 5 Wood units (WU) or ≥ 400 dyn·sec·cm-5 and a pulmonary artery wedge pressure (PAWP) of ≤ 15 mm Hg.
4. Diagnosis of WHO pulmonary arterial hypertension (PAH) Group 1.
5. Symptomatic PAH classified as WHO Functional class II to IV.
6. On stable doses of at least 2 approved background PAH therapies and diuretics for at least 90 days prior to Screening.
7. 6-Minute Walk Distance (6MWD) ≥ 150m and ≤ 500m repeated twice during screening.
8. Ability to adhere to study visit schedule and understand and comply with all protocol requirements.

Exclusion Criteria:

1. Hospitalization for any worsening medical condition or major surgery within 4 weeks prior to screening.
2. Any symptomatic coronary disease events within 6 months of the screening visit.
3. History of heart transplant or on heart transplant list.
4. Uncontrolled systemic hypertension.
5. History of restrictive, constrictive or congestive cardiomyopathy.
6. History of significant valvular stenosis or regurgitation.
7. Untreated or poorly controlled moderate or severe obstructive sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Number of Adverse Events (AEs) | up to 24 weeks
  An AE is any untoward medical occurrence in a patient or clinical trial patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The incidence and number of patients who experience an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Champagne, M.Sc, Study Director — 35Pharma Inc